CLINICAL TRIAL: NCT00167674
Title: ARVs to Prevent Breastmilk HIV:Viral and Immune Responses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-5529-A03; Elizabeth Glaser (Other Grant/Funding Number: Scientist Award #11-03)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: breastmilk; HIV-1; antiretroviral; mother-to-child; transmission
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): Combined short-course Zidovudine/Nevirapine
  Interventions: Drug: Combined short-course zidovudine/nevirapine
- A (Experimental): HAART during pregnancy and 6 months postpartum
  Interventions: Drug: HAART

INTERVENTIONS:
Drug: Combined short-course zidovudine/nevirapine — 300 mg of ZDV was given twice daily from 34 weeks gestation until labor then every 3 hours until delivery; 200 mg of NVP was given as a single oral dose at the onset of labor; and a single 2 mg/kg (6 mg if birthweight > 2.5 kg) oral dose of NVP suspension was administered to the infant within 72 hours of delivery.
  Arms: B
Drug: HAART — 300 mg of zidovudine (ZDV), 150 mg of lamivudine, and 200 mg nevirapine (NVP) was given twice daily from 34 weeks gestation until six months after delivery.
  Arms: A

SUMMARY:
Identifying new approaches for preventing breastmilk transmission of HIV-1 is an important research priority. To this end, clinical trials are underway to evaluate the efficacy of HAART (zidovudine, lamivudine, nevirapine) during late pregnancy/lactation versus zidovudine/nevirapine peripartum for prevention of breastmilk HIV-1 transmission. It is important to understand the mechanism of effect of these antiretroviral (ARV) strategies on prevention of breastmilk HIV-1 transmission.

This phase II trial will compare HAART vs peripartum zidovudine/nevirapine for effect on breastmilk HIV-1, breastmilk HIV-1 specific immune responses, and infant HIV-1 specific immune responses.

100 pregnant HIV-1 seropositive women in Nairobi with CD4 counts between 200 to 500 who have chosen to breastfeed will receive either ARV regimen. Mother-infant pairs will be followed for 1 year after delivery. Home visits will be conducted in the first month (~10 visits) to collect 2-5 mls of breastmilk per visit. Mother-infant pairs will be seen in the study clinic with maternal blood and breastmilk and infant blood collected at months 1, 3, and 6 for HIV-1 and HIV-1 Elispot assays. Breastmilk HIV-1 RNA and DNA levels will be quantified in Dr. Overbaugh's laboratory in Seattle and Elispot assays conducted in Nairobi with validation of a subset in Dr. Rowland-Jones laboratory in Oxford. Viral loads, decay curves, half-life, and re-population following ARV cessation will be estimated for each regimen and regimens compared. These studies will provide insight into the viral and immune responses to ARV regimens proposed for prevention of breastfeeding HIV-1 transmission and will be important for rational design of future interventions. After taking into account, estimated loss to follow-up, the targeted sample size with outcome data was 80 women, 40 in each trial arm, estimating undetectable breast milk HIV-1 RNA levels in the HAART arm and median breast milk HIV-1 RNA levels of 3.0 log10 in women receiving ZDV/NVP.

DETAILED DESCRIPTION:
This will be a randomized study comparing breastfeeding women receiving zidovudine/nevirapine (from 36 weeks to delivery/first day postpartum) to women receiving HAART (zidovudine, nevirapine, lamivudine) initiated at 36 weeks and continuing throughout lactation (recommended for 6 months, breastfeeding cessation prior to HAART cessation).

This a prospective cohort study that will follow HIV-1 seropositive women and their infants to be conducted in Nairobi. Women with CD4 counts between 200 and 500 will be randomized to one of the two regimens and compared.

The study procedures are outlined below:

1. Voluntary HIV-1 counseling and testing in a Nairobi City council antenatal clinic: collection of blood using venipuncture following written informed consent.
2. Enrollment of HIV-1 infected women into new cohort before 32 wks gestation after written informed consent
3. Routine antenatal care including STD screening and multivitamins/iron
4. Collection of maternal blood and genital specimens at 32 weeks for STD diagnosis, HIV-1 RNA levels, CD4 counts, liver function tests, and complete blood counts.
5. Assignment to treatment depending on CD4 count at 34 weeks:

   1. CD4>500 zidovudine/nevirapine short-course treatment
   2. CD4 200-500 randomization to zidovudine/nevirapine short-course or 3-drugs (nevirapine, zidovudine, and 3TC) during pregnancy and breastfeeding, with recommendation to stop breastfeeding at 6 months and the drugs to stop after cessation of breastfeeding
   3. CD4<200 3-drug regimen (nevirapine, zidovudine, and 3TC) through pregnancy and breastfeeding continued after cessation of breastfeeding with referral to sites in Nairobi providing long-term treatment
6. At delivery collection of maternal breastmilk (2-5 mls), cord blood (15 mls), maternal blood (15 mls), and infant blood (3 mls) for HIV-1 RNA, CD4 counts, HIV-1 specific CTL assays, complete blood counts, and liver function tests.
7. Collection of maternal breastmilk (2-5 mls) from home visits 3 times per week in the first 2 weeks, then 2 times per week for the next two weeks. Filter paper blood specimens will be collected weekly at the home visits.
8. Women receiving the 3-drug regimen who have expressible breastmilk after cessation of breastfeeding and cessation of drugs will also have home collection (3-5 mls) of specimens 3-times weekly for 2 weeks after cessation of breastfeeding.
9. Clinic visits at week 2, month 1, 3, and 6 with breastmilk and blood collection. Higher volumes of breastmilk (~25 -50 mls) will be collected at the clinic visits (w2, m1, 3, and 6) for HIV-1 RNA, DNA and HIV-1 specific immune assays. Collection of maternal blood at week 2, month 1, 3, and 6 for HIV-1 RNA levels, CD4 counts, HIV-1 CTL levels, liver function tests, and complete blood counts.
10. Collection of infant blood at m1, 3, and 6 for HIV-1 and HIV-1 specific immune responses. Heel prick filter paper assays at months 9 and 12 for HIV-1 DNA PCR assays.

ELIGIBILITY:
Inclusion Criteria:

* The subject population is recruited from Mathare North Clinic in Nairobi, Kenya where voluntary HIV-1 counseling and testing is offered to pregnant women
* Pregnant women who test positive for HIV-1 antibody are eligible for the study if they are over 18 years of age
* At less than 32 weeks' gestation
* Have never previously been exposed to antiretroviral medications
* Agree to serial maternal blood
* Breast milk
* Infant blood draws
* Plan to live in Nairobi for at least a year after delivery.

Exclusion Criteria:

* CD4 >500 or <200
* Not planning to live in Nairobi after delivery
* Not planning to breastfeed.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2003-11-03 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace C. John-Stewart, MD, PhD, Principal Investigator — University of Washington; Carey Farquhar, MD, MPH, Study Director — University of Washington; Dorothy Mbori-Ngacha, MBChB,MPH, Study Director — University of Nairobi; Ruth Nduati, MBChB,MPH, Study Director — University of Nairobi; James Kiarie, MBChB, MPH, Study Director — University of Nairobi; Michael Chung, MD, MPH, Study Director — University of Washington; Julie Overbaugh, PhD, Study Director — Fred Hutchinson Cancer Center; John Kinuthia, MBChB, MMed, Study Director — University of Nairobi; Barbra Richardson, PhD, Study Director — University of Washington
Locations (1):
- University of Nairobi, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
may request data from PI

REFERENCES:
- [Background] Chung MH, Kiarie JN, Richardson BA, Lehman DA, Overbaugh J, Njiri F, John-Stewart GC. Independent effects of nevirapine prophylaxis and HIV-1 RNA suppression in breast milk on early perinatal HIV-1 transmission. J Acquir Immune Defic Syndr. 2007 Dec 1;46(4):472-8. doi: 10.1097/qai.0b013e3181594c1c. PMID 18077838
- [Result] Lehman DA, Chung MH, John-Stewart GC, Richardson BA, Kiarie J, Kinuthia J, Overbaugh J. HIV-1 persists in breast milk cells despite antiretroviral treatment to prevent mother-to-child transmission. AIDS. 2008 Jul 31;22(12):1475-85. doi: 10.1097/QAD.0b013e328302cc11. PMID 18614871
- [Result] Chung MH, Kiarie JN, Richardson BA, Lehman DA, Overbaugh J, Kinuthia J, Njiri F, John-Stewart GC. Highly active antiretroviral therapy versus zidovudine/nevirapine effects on early breast milk HIV type-1 Rna: a phase II randomized clinical trial. Antivir Ther. 2008;13(6):799-807. PMID 18839781
- [Result] Lehman DA, Chung MH, Mabuka JM, John-Stewart GC, Kiarie J, Kinuthia J, Overbaugh J. Lower risk of resistance after short-course HAART compared with zidovudine/single-dose nevirapine used for prevention of HIV-1 mother-to-child transmission. J Acquir Immune Defic Syndr. 2009 Aug 15;51(5):522-9. doi: 10.1097/QAI.0b013e3181aa8a22. PMID 19502990
- [Derived] Slyker JA, Richardson B, Chung MH, Atkinson C, Asbjornsdottir KH, Lehman DA, Boeckh M, Emery V, Kiarie J, John-Stewart G. Maternal Highly Active Antiretroviral Therapy Reduces Vertical Cytomegalovirus Transmission But Does Not Reduce Breast Milk Cytomegalovirus Levels. AIDS Res Hum Retroviruses. 2017 Apr;33(4):332-338. doi: 10.1089/AID.2016.0121. Epub 2016 Dec 6. PMID 27796131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment between Nov 3, 2003 and Mar 11, 2005 Mathare North City Council Clinic
Groups:
- ZDV/NVP: Combined short-course Zidovudine/Nevirapine
  Combined short-course zidovudine/nevirapine: 300 mg of ZDV was given twice daily from 34 weeks gestation until labor then every 3 hours until delivery; 200 mg of NVP was given as a single oral dose at the onset of labor; and a single 2 mg/kg (6 mg if birthweight > 2.5 kg) oral dose of NVP suspension was administered to the infant within 72 hours of delivery.
- HAART: HAART during pregnancy and 6 months postpartum
  HAART: 300 mg of zidovudine (ZDV), 150 mg of lamivudine, and 200 mg nevirapine (NVP) was given twice daily from 34 weeks gestation until six months after delivery.
Period: Overall Study
Arm/Group | ZDV/NVP | HAART
Started | 28 | 30
Completed | 24 | 24
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZDV/NVP | HAART | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [20 to 31] | 26 [24 to 29] | 25 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 28 | 30 | 58
  Africa | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Outcome 1: Serial HIV-1 RNA Levels in Breastmilk.
Time Frame: Weeks 0, 1, 2, 3 and 4
Population: Participants with VL data available.
Measure: Median (Inter-Quartile Range); unit: Log10 Viral load copies/ml
Arm/Group | ZDV/NVP | HAART
Number analyzed (Participants) | 24 | 26
Log10 Viral load copies/ml
  Week 0: number analyzed (Participants) | 12 | 11
  Week 0 | 2.74 [2.23 to 3.43] | 2.03 [1.70 to 2.41]
  Week 1: number analyzed (Participants) | 22 | 26
  Week 1 | 1.70 [1.70 to 2.35] | 1.70 [1.70 to 1.73]
  Week 2 | 1.70 [1.70 to 2.14] | 1.70 [1.70 to 1.70]
  Week 3 | 2.22 [1.91 to 3.12] | 1.70 [1.70 to 1.70]
  Week 4: number analyzed (Participants) | 24 | 25
  Week 4 | 2.11 [1.70 to 3.07] | 1.70 [1.70 to 1.70]

ADVERSE EVENTS:
Arm/Group | ZDV/NVP | HAART
All-Cause Mortality (participants affected / at risk) | 3/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 3/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZDV/NVP (N=24) | HAART (N=26)
Death (Infections and infestations) | 3 (3) | 0 (0) — Mortality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No